CLINICAL TRIAL: NCT06268964
Title: Comparative Effect of Trimebutine and Probiotics on Functional Abdominal Pain Disorders (FAPD) in Children: Randomized Clinical Trial (RCT)
Brief Title: Exploring Treatments for Children's Abdominal Pain: Comparing Trimebutine and Probiotics
Acronym: FAPD_RCT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universidad de Colima (Other)
Responsible Party: Principal Investigator, Fabian Rojas Larios, Doctor of Science, Universidad de Colima
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-5
Record Dates: First submitted 2024-01-23; First posted 2024-02-21 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Functional Abdominal Pain Syndrome; Functional Gastrointestinal Disorders; Irritable Bowel Syndrome Variant of Childhood
Keywords: functional abdominal pain; randomized clinical trial; placebo; double-blind; trimebutine; Lactobacillus rhamnosus; pediatrics
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Trimebutine; microcrystalline cellulose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trimebutine + Probiotic (Experimental): Participants received trimebutine in 200 mg tablets or 20 mg/ml suspension at a dose of 15 mg/kg/day adjusted to their weight, divided into 2 doses (morning and night) + Lactobacillus rhamnosus 5 billion Colony Forming Units (CFUs) in chewable tablets, a single dose (night), for a period of 8 weeks.
  Interventions: Drug: Trimebutine; Dietary Supplement: Lactobacillus rhamnosus
- Trimebutine + Placebo (Active Comparator): Participants received trimebutine in 200 mg tablets or 20 mg/ml suspension at a dose of 15 mg/kg/day adjusted to their weight, divided into 2 doses (morning and night) + Placebo, 250 mg microcrystalline cellulose tablets, a single dose (night), for a period of 8 weeks.
  Interventions: Drug: Trimebutine; Other: Placebo
- Probiotic + Placebo (Active Comparator): Participants received Lactobacillus rhamnosus 5 billion Colony Forming Units (CFUs) in chewable tablets + Placebo, 250 mg microcrystalline cellulose tablets, a single dose (night), for a period of 8 weeks.
  Interventions: Dietary Supplement: Lactobacillus rhamnosus; Other: Placebo

INTERVENTIONS:
Drug: Trimebutine — Prescription of trimebutine at pediatric dosage (15 mg/kg/day), divided into 2 daily doses, for 8 weeks.
  Arms: Trimebutine + Placebo; Trimebutine + Probiotic
Dietary Supplement: Lactobacillus rhamnosus — Prescription of Lactobacillus rhamnosus 5 billion CFUs in chewable tablets, a single dose (night) for 8 weeks.
  Arms: Probiotic + Placebo; Trimebutine + Probiotic
Other: Placebo — Prescription of a placebo, 250 mg microcrystalline cellulose tablets, a single dose (night) for 8 weeks.
  Other Names: Microcrystalline cellulose
  Arms: Probiotic + Placebo; Trimebutine + Placebo

SUMMARY:
The goal of this clinical trial is to test the effectiveness of trimebutine and probiotics in treating Functional Abdominal Pain Disorders (FAPD) in a pediatric population. The main questions it aims to answer are: Is trimebutine effective in reducing the symptoms of FAPD in children? Are probiotics effective in reducing the symptoms of FAPD in children? Participants will be randomly assigned to one of three treatment groups (trimebutine/probiotics, probiotics/placebo, or trimebutine/placebo). Undergo measurements for pain and other relevant metrics at the start of the study, after 4 weeks, and after 8 weeks.

Researchers will compare the trimebutine/probiotics group to the probiotics/placebo and the trimebutine/placebo groups to see if there are significant differences in the efficacy of these treatments in reducing symptoms of FAPD in children.

DETAILED DESCRIPTION:
The protocol will be submitted for review by the Research Committee and the Ethics Committee of the Regional University Hospital of Colima. Upon receiving approval, a double-blind, placebo-controlled, randomized clinical trial will be carried out, based on CONSORT guidelines. This trial involves the participation of pediatric patients aged 4 to 18.

Patients will be selected from those attending private practice and satisfying Rome IV criteria for any of the Functional Abdominal Pain Disorders (FAPD). Before any intervention takes place, the purpose and procedures of the study will be explained to both the patients and their legal guardians. If they decide to participate, they will be asked to sign an informed consent letter and assent form for minors. Patients will be selected through stratified probabilistic sampling in 4 categories (Irritable Bowel Syndrome, Functional Dyspepsia, Abdominal Migraine, and Functional Abdominal Pain not otherwise specified (FAP-NOS)) until the desired sample size of 82 participants is reached. Once participants are selected, they will be randomly assigned to one of the three groups: trimebutine/probiotic, probiotic/placebo, or trimebutine/placebo, with each group consisting of at least 20 participants. The initial diagnosis will be carried out using the Rome IV Criteria Questionnaires for pediatric patients, and the intensity of pain will be evaluated using the Visual Analog Scale (VAS) and quality of life with PedsQL 4.0. Patients will be administered the treatment corresponding to their assigned group and will be clinically followed up at 4 and 8 weeks. During these follow-up consultations, the Rome IV Criteria Questionnaires and scales will be reapplied to assess the evolution of the patients' symptoms and their response to treatment. Any patient who requests voluntary withdrawal, those with treatment adherence less than 80%, and those participating in another study or being treated by another physician simultaneously will be removed from the study.

Statistical analysis will be carried out using international Business Machine (IBM®) Statistical Package for the Social Sciences (SPSS®) Statistics 26. Descriptive statistics with measures of central tendency will be used, presenting the results in tables and graphs. To determine whether the data follow a normal distribution, the Kolmogorov-Smirnov and Shapiro-Wilk tests will be applied. Measurements in 3 groups (trimebutine, probiotics, and control) and at 3 times (0, 4, and 8 weeks) will be analyzed. For intervening categorical variables like gender and education, the chi-square test (X2) will be used. For continuous variables like age and BMI, the Mann-Whitney U test will be applied, expecting statistically significant differences with p < 0.05.

If the data follow a normal distribution, repeated measures ANOVA will be used to compare the means of the 3 groups (trimebutine, probiotics, and placebo). McNemar's test or the sign test will be considered as secondary analyses to evaluate changes within each group over time (0, 4, and 8 weeks). If the data do not follow a normal distribution, non-parametric tests like the Friedman test will be employed.

In case of finding a statistically significant difference in repeated measures ANOVA or the Friedman test, post hoc tests will be performed to identify specific differences between groups and times. If necessary, correlation tests like Pearson or Spearman will be used to evaluate relationships between different variables within the study.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients from 4 to 18 years old.
* Meeting the Rome IV criteria for any of the Functional Abdominal Pain Disorders (Functional Dyspepsia, Irritable Bowel Syndrome, Abdominal Migraine or Functional Abdominal Pain Not Otherwise Specified)
* Having the informed consent signed by the parents or legal guardians of the minor.

Exclusion Criteria:

* Patients presenting abdominal pain of organic cause.
* Immunosuppressed patients.
* Patients with previous hypersensitivity to the study drug.

Elimination Criteria:

* Voluntary withdrawal from the study.
* Patients not adhering to treatment (less than 80%)
* Patients participating in another study simultaneously.
* Patients being treated by another doctor simultaneously.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 82 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Average Score on Visual Analog Scale for Abdominal Pain | Baseline to 8 weeks post-treatment.
  Participants rated the highest intensity of abdominal pain they experienced during the past eight weeks on a scale of 0 (no pain) to 10 (worst pain imaginable), using an Visual Analog Scale (VAS) scale. A decrease in the score signifies an improvement in symptoms.

SECONDARY OUTCOMES:
Improvement in Quality of Life with PedsQL 3.0 | Baseline to 8 weeks post-treatment.
  Impact of the treatment on the Quality of Life in pediatric patients with FAPD. The PedsQL 0 - 100 scoring system is used, where higher scores indicate better quality of life. The change in scores from baseline to 8 weeks post-treatment is measured.
Improvement in Quality of Life with PedsQL 3.0 | Baseline to 4 weeks post-treatment.
  Impact of the treatment on the Quality of Life in pediatric patients with FAPD. The PedsQL 0 - 100 scoring system is used, where higher scores indicate better quality of life. The change in scores from baseline to 4 weeks post-treatment is measured.
Average Score on Visual Analog Scale for Abdominal Pain | Baseline to 4 weeks post-treatment.
  Participants rated the highest intensity of abdominal pain they experienced during the past eight weeks on a scale of 0 (no pain) to 10 (worst pain imaginable), using an Visual Analog Scale (VAS) scale. A decrease in the score signifies an improvement in symptoms.

OTHER OUTCOMES:
Number of Participants with Treatment-Related Adverse Events | Baseline to 8 weeks post-treatment.
  Number and type of treatment-related adverse events reported during the study period, evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo H Sandoval-Villaseñor, MD, Principal Investigator — Universidad de Colima; Fabián Rojas-Larios, PhD, Study Director — Universidad de Colima; Carmen A Sánchez-Ramírez, PhD, Study Director — Universidad de Colima
Locations (1):
- School of Medicine, University of Colima, Colima, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Korterink JJ, Diederen K, Benninga MA, Tabbers MM. Epidemiology of pediatric functional abdominal pain disorders: a meta-analysis. PLoS One. 2015 May 20;10(5):e0126982. doi: 10.1371/journal.pone.0126982. eCollection 2015. PMID 25992621
- [Background] Simren M, Tornblom H, Palsson OS, Van Oudenhove L, Whitehead WE, Tack J. Cumulative Effects of Psychologic Distress, Visceral Hypersensitivity, and Abnormal Transit on Patient-reported Outcomes in Irritable Bowel Syndrome. Gastroenterology. 2019 Aug;157(2):391-402.e2. doi: 10.1053/j.gastro.2019.04.019. Epub 2019 Apr 22. PMID 31022401
- [Background] Thapar N, Benninga MA, Crowell MD, Di Lorenzo C, Mack I, Nurko S, Saps M, Shulman RJ, Szajewska H, van Tilburg MAL, Enck P. Paediatric functional abdominal pain disorders. Nat Rev Dis Primers. 2020 Nov 5;6(1):89. doi: 10.1038/s41572-020-00222-5. PMID 33154368
- [Background] Ding FCL, Karkhaneh M, Zorzela L, Jou H, Vohra S. Probiotics for paediatric functional abdominal pain disorders: A rapid review. Paediatr Child Health. 2019 Sep;24(6):383-394. doi: 10.1093/pch/pxz036. Epub 2019 May 4. PMID 31528110
- [Background] Horvath A, Dziechciarz P, Szajewska H. Systematic review of randomized controlled trials: fiber supplements for abdominal pain-related functional gastrointestinal disorders in childhood. Ann Nutr Metab. 2012;61(2):95-101. doi: 10.1159/000338965. PMID 22889919
- [Background] Chumpitazi BP, Kearns GL, Shulman RJ. Review article: the physiological effects and safety of peppermint oil and its efficacy in irritable bowel syndrome and other functional disorders. Aliment Pharmacol Ther. 2018 Mar;47(6):738-752. doi: 10.1111/apt.14519. Epub 2018 Jan 26. PMID 29372567
- [Background] Karabulut GS, Beser OF, Erginoz E, Kutlu T, Cokugras FC, Erkan T. The Incidence of Irritable Bowel Syndrome in Children Using the Rome III Criteria and the Effect of Trimebutine Treatment. J Neurogastroenterol Motil. 2013 Jan;19(1):90-3. doi: 10.5056/jnm.2013.19.1.90. Epub 2013 Jan 8. PMID 23350053
- [Background] Wallace C, Gordon M, Sinopoulou V, Akobeng AK. Probiotics for management of functional abdominal pain disorders in children. Cochrane Database Syst Rev. 2023 Feb 17;2(2):CD012849. doi: 10.1002/14651858.CD012849.pub2. PMID 36799531
- [Background] Hyams JS, Di Lorenzo C, Saps M, Shulman RJ, Staiano A, van Tilburg M. Functional Disorders: Children and Adolescents. Gastroenterology. 2016 Feb 15:S0016-5085(16)00181-5. doi: 10.1053/j.gastro.2016.02.015. Online ahead of print. PMID 27144632
- [Background] Khrizman M, Pakalnis A. Management of Pediatric Migraine: Current Therapies. Pediatr Ann. 2018 Feb 1;47(2):e55-e60. doi: 10.3928/19382359-20180129-02. PMID 29446795
- [Background] Saps M, Velasco-Benitez CA, Langshaw AH, Ramirez-Hernandez CR. Prevalence of Functional Gastrointestinal Disorders in Children and Adolescents: Comparison Between Rome III and Rome IV Criteria. J Pediatr. 2018 Aug;199:212-216. doi: 10.1016/j.jpeds.2018.03.037. Epub 2018 May 7. PMID 29747935
- [Background] Koppen IJ, Nurko S, Saps M, Di Lorenzo C, Benninga MA. The pediatric Rome IV criteria: what's new? Expert Rev Gastroenterol Hepatol. 2017 Mar;11(3):193-201. doi: 10.1080/17474124.2017.1282820. Epub 2017 Jan 24. PMID 28092724
- [Background] Chiou E, Nurko S. Management of functional abdominal pain and irritable bowel syndrome in children and adolescents. Expert Rev Gastroenterol Hepatol. 2010 Jun;4(3):293-304. doi: 10.1586/egh.10.28. PMID 20528117
- [Background] Koppen IJN, Saps M, Lavigne JV, Nurko S, Taminiau JAJM, Di Lorenzo C, Benninga MA. Recommendations for pharmacological clinical trials in children with functional constipation: The Rome foundation pediatric subcommittee on clinical trials. Neurogastroenterol Motil. 2018 Apr;30(4):e13294. doi: 10.1111/nmo.13294. Epub 2018 Jan 30. PMID 29380480
- [Background] Benninga MA, Faure C, Hyman PE, St James Roberts I, Schechter NL, Nurko S. Childhood Functional Gastrointestinal Disorders: Neonate/Toddler. Gastroenterology. 2016 Feb 15:S0016-5085(16)00182-7. doi: 10.1053/j.gastro.2016.02.016. Online ahead of print. PMID 27144631
- [Background] Devanarayana NM, Rajindrajith S. Irritable bowel syndrome in children: Current knowledge, challenges and opportunities. World J Gastroenterol. 2018 Jun 7;24(21):2211-2235. doi: 10.3748/wjg.v24.i21.2211. PMID 29881232
- [Background] van Tilburg MA, Hyman PE, Walker L, Rouster A, Palsson OS, Kim SM, Whitehead WE. Prevalence of functional gastrointestinal disorders in infants and toddlers. J Pediatr. 2015 Mar;166(3):684-9. doi: 10.1016/j.jpeds.2014.11.039. Epub 2014 Dec 31. PMID 25557967
- [Background] Chumpitazi BP, Weidler EM, Lu DY, Tsai CM, Shulman RJ. Self-Perceived Food Intolerances Are Common and Associated with Clinical Severity in Childhood Irritable Bowel Syndrome. J Acad Nutr Diet. 2016 Sep;116(9):1458-1464. doi: 10.1016/j.jand.2016.04.017. Epub 2016 Jun 15. PMID 27316779
- [Background] Van Oudenhove L, Crowell MD, Drossman DA, Halpert AD, Keefer L, Lackner JM, Murphy TB, Naliboff BD, Levy RL. Biopsychosocial Aspects of Functional Gastrointestinal Disorders. Gastroenterology. 2016 Feb 18:S0016-5085(16)00218-3. doi: 10.1053/j.gastro.2016.02.027. Online ahead of print. PMID 27144624
- [Background] Halmos EP, Power VA, Shepherd SJ, Gibson PR, Muir JG. A diet low in FODMAPs reduces symptoms of irritable bowel syndrome. Gastroenterology. 2014 Jan;146(1):67-75.e5. doi: 10.1053/j.gastro.2013.09.046. Epub 2013 Sep 25. PMID 24076059
- [Background] Newlove-Delgado TV, Martin AE, Abbott RA, Bethel A, Thompson-Coon J, Whear R, Logan S. Dietary interventions for recurrent abdominal pain in childhood. Cochrane Database Syst Rev. 2017 Mar 23;3(3):CD010972. doi: 10.1002/14651858.CD010972.pub2. PMID 28334433
- [Background] Ford AC, Quigley EM, Lacy BE, Lembo AJ, Saito YA, Schiller LR, Soffer EE, Spiegel BM, Moayyedi P. Efficacy of prebiotics, probiotics, and synbiotics in irritable bowel syndrome and chronic idiopathic constipation: systematic review and meta-analysis. Am J Gastroenterol. 2014 Oct;109(10):1547-61; quiz 1546, 1562. doi: 10.1038/ajg.2014.202. Epub 2014 Jul 29. PMID 25070051
- [Background] Chumpitazi BP, Cope JL, Hollister EB, Tsai CM, McMeans AR, Luna RA, Versalovic J, Shulman RJ. Randomised clinical trial: gut microbiome biomarkers are associated with clinical response to a low FODMAP diet in children with the irritable bowel syndrome. Aliment Pharmacol Ther. 2015 Aug;42(4):418-27. doi: 10.1111/apt.13286. Epub 2015 Jun 24. PMID 26104013
- [Background] Rutten JM, Reitsma JB, Vlieger AM, Benninga MA. Gut-directed hypnotherapy for functional abdominal pain or irritable bowel syndrome in children: a systematic review. Arch Dis Child. 2013 Apr;98(4):252-7. doi: 10.1136/archdischild-2012-302906. Epub 2012 Dec 6. PMID 23220208
- [Background] Palsson OS, Whitehead WE. Psychological treatments in functional gastrointestinal disorders: a primer for the gastroenterologist. Clin Gastroenterol Hepatol. 2013 Mar;11(3):208-16; quiz e22-3. doi: 10.1016/j.cgh.2012.10.031. Epub 2012 Oct 24. PMID 23103907
- [Background] Kountouras J, Gavalas E, Papaefthymiou A, Tsechelidis I, Polyzos SA, Bor S, Diculescu M, Jadallah Kappa, Tadeusz M, Karakan T, Bochenek Alpha, Rozciecha J, Dabrowski P, Sparchez Z, Sezgin O, Gulten M, Farsakh NA, Doulberis M. Trimebutine Maleate Monotherapy for Functional Dyspepsia: A Multicenter, Randomized, Double-Blind Placebo Controlled Prospective Trial. Medicina (Kaunas). 2020 Jul 8;56(7):339. doi: 10.3390/medicina56070339. PMID 32650518
- [Background] Vandenplas Y, Hauser B, Salvatore S. Functional Gastrointestinal Disorders in Infancy: Impact on the Health of the Infant and Family. Pediatr Gastroenterol Hepatol Nutr. 2019 May;22(3):207-216. doi: 10.5223/pghn.2019.22.3.207. Epub 2019 Apr 16. PMID 31110953
- [Background] Salminen S, Collado MC, Endo A, Hill C, Lebeer S, Quigley EMM, Sanders ME, Shamir R, Swann JR, Szajewska H, Vinderola G. The International Scientific Association of Probiotics and Prebiotics (ISAPP) consensus statement on the definition and scope of postbiotics. Nat Rev Gastroenterol Hepatol. 2021 Sep;18(9):649-667. doi: 10.1038/s41575-021-00440-6. Epub 2021 May 4. PMID 33948025
- [Background] Dryl R, Szajewska H. Probiotics for management of infantile colic: a systematic review of randomized controlled trials. Arch Med Sci. 2018 Aug;14(5):1137-1143. doi: 10.5114/aoms.2017.66055. Epub 2017 Feb 16. PMID 30154898
- [Background] Francavilla R, Miniello V, Magista AM, De Canio A, Bucci N, Gagliardi F, Lionetti E, Castellaneta S, Polimeno L, Peccarisi L, Indrio F, Cavallo L. A randomized controlled trial of Lactobacillus GG in children with functional abdominal pain. Pediatrics. 2010 Dec;126(6):e1445-52. doi: 10.1542/peds.2010-0467. Epub 2010 Nov 15. PMID 21078735
- [Background] Romano C, Ferrau' V, Cavataio F, Iacono G, Spina M, Lionetti E, Comisi F, Famiani A, Comito D. Lactobacillus reuteri in children with functional abdominal pain (FAP). J Paediatr Child Health. 2014 Oct;50(10):E68-71. doi: 10.1111/j.1440-1754.2010.01797.x. Epub 2010 Jul 8. PMID 20626584
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; CONSORT. CONSORT 2010 explanation and elaboration: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2012;10(1):28-55. doi: 10.1016/j.ijsu.2011.10.001. Epub 2011 Oct 12. PMID 22036893

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-01-09): https://cdn.clinicaltrials.gov/large-docs/64/NCT06268964/Prot_SAP_ICF_000.pdf